CLINICAL TRIAL: NCT01150201
Title: Phase 4 Study of the Renoprotective Efficacy of Aliskiren in Addition to Angiotensin II Receptor Blocker in Chronic Kidney Disease
Brief Title: Aliskiren Combined With Losartan in Proteinuric, Non-diabetic Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sydney C.W. TANG/ Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Novartis-ST-02
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Kidney Disease
Keywords: CKD; proteinuria; eGFR; Progression of chronic kidney disease
MeSH Terms: conditions — Kidney Diseases; Proteinuria | interventions — aliskiren; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Experimental): Aliskiren
  Interventions: Drug: Aliskiren
- Losartan (Active Comparator): ARB
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Aliskiren — For CKD treatment
  Other Names: Rasilez
  Arms: Aliskiren
Drug: Losartan — Control
  Other Names: Cozaar
  Arms: Losartan

SUMMARY:
Study objective: To investigate the potential anti-proteinuric and renoprotective efficacy of aliskiren in addition to losartan in patients at risk of developing end-stage renal disease (ESRD)

Methods: This will be a randomized, double-blind study in which proteinuric, non-diabetic patients with chronic kidney disease (CKD) will be assigned in a 1:1 ratio to one of the following treatment groups for 3 years:

* Group A: Losartan (Control arm: conventional treatment)*
* Group B: Aliskiren plus Losartan (Intervention arm)*

  * With optional addition of other anti-hypertensive agents to achieve an optimal target blood pressure of <130/80 mmHg.

DETAILED DESCRIPTION:
Aliskiren is a direct renin inhibitor that has been shown to reduce proteinuria and retard renal deterioration in type 2 diabetic patients with overt nephropathy. However, it is not known if these therapeutic effects can be extended to nondiabetic chronic renal disease. The current study aims to explore this research question by randomly assigning patients with various stages of chronic renal disease to receive either aliskiren on top of losartan, or continuation of losartan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 - 80 years of age
* Presence of nondiabetic CKD stages 3 to 4 as defined by estimated glomerular filtration rate (eGFR by 4-variable MDRD equation) as follows:

  * Stage 3: Moderate decrease in GFR 30-59 mL/min/1.73 sq.m
  * Stage 4: Severe decrease in GFR 15-29 mL/min/1.73 sq.m
  * CKD is defined as either kidney damage or GFR <60 mL/min/1.73 m2 for > 3 months with variations of less than 30% in the 3 months before screening
* Early-morning urinary protein-to-creatinine ratio of >500 mg/g or 57 mg/mmol on at least 2 occasions four weeks apart
* Patients who are willing to give written, informed consent

Exclusion Criteria:

* eGFR < 15 or > 60 ml/min/1.73m2
* Early-morning urinary protein-to-creatinine ratio of >5000 mg/g or 570 mg/mmol, or urinary protein-to-creatinine ratio of <500 mg/g or 57 mg/mmol
* Serum K+ > 5.2 mmol/L
* Presence of bilateral renal artery stenosis
* Known allergy to losartan or aliskiren
* Patients who are receiving angiotensin II receptor blocker / angiotensin converting enzyme inhibitor combination within 12 weeks of randomization
* Concurrent treatment with corticosteroids, nonsteroidal antiinflammatory drugs, or immunosuppressive agent
* Patients with connective tissue disease or obstructive uropathy
* Patients with concomitant malignancy or any such conditions that will severely limit life expectancy
* Female who are pregnant or intending to conceive
* Female of child-bearing age who are unwilling to practice effective contraception
* Patients who are unable to give informed consent
* Patients simultaneously participating in another study or who have participated in another study within the last 30 days of entry into this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Rate of change in GFR | 36 months

SECONDARY OUTCOMES:
Change in proteinuria | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Sydney CW Tang, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China